CLINICAL TRIAL: NCT00137254
Title: Effects of Insulin on Post Burn Hypermetabolism
Brief Title: Insulin on Post Burn Hypermetabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Collaborators: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-05-004; NIH RO-1 GM063120-02
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Burns
Keywords: Severe burns; Hyperinsulinemia; Insulin; Muscle protein kinetics; Immune function; Exercise
MeSH Terms: conditions — Burns; Hyperinsulinism; Insulin Resistance; Motor Activity | interventions — Insulin; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator)
  Interventions: Drug: Insulin; Drug: Stable Isotopes; Drug: Indocyanine Green

INTERVENTIONS:
Drug: Insulin — IV insulin
Drug: Stable Isotopes — IV administration of stable isotopes
Drug: Indocyanine Green — IV administration of ICG

SUMMARY:
The purpose of this study is to examine the effects of insulin on helping burn patients recover faster from their burns.

DETAILED DESCRIPTION:
Severe injuries produce profound hypermetabolic stress responses which cause severe loss of lean body mass and muscle wasting, immunologic compromise, slowed wound healing, and related bone loss, all which contribute to increased morbidity, mortality, and prolonged recovery from injury. The results of hypermetabolism persist for weeks to months depending on the severity of the insult. Massive burns can cause severe catabolism and are an excellent model to study the general effects of injury on protein metabolism. Severe burns are characterized by dramatic increases in energy utilization and alterations in the metabolism of carbohydrates, fat, and protein.

Insulin treatment improves net protein synthesis in the severely burned, principally through improved muscle protein synthesis. Although controversy exist as to whether insulin is effective as an anabolic hormone through increasing protein synthesis or decreasing protein breakdown, we believe that consideration of the methods and experimental protocols used in the various studies bear consideration when evaluating this topic.

ELIGIBILITY:
Inclusion Criteria:

* Burn equal to or greater than 20% total body surface area (TBSA)
* Between the ages of 18-72 years
* Burns occurred within 14 days of coming to burn center

Exclusion Criteria:

* Heart attack within 3 months
* Have or have had cancer
* Seizure disorder
* Pregnancy
* Pre-existing arterial insufficiency
* Diabetes or known history of hypoglycemia
* Allergy to iodine or shellfish

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To determine the effect of euglycemic hyperinsulinemia throughout the hospital course on net muscle protein synthesis, and to relate continued muscle anabolism to improved lean body mass and improved functional recovery in severely burned patients | 45 days
To assess the relationship of insulin physiologic and molecular effects on skeletal muscle in severely burned patients | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Wolf, MD, Principal Investigator — US Army Institute of Surgical Research
Locations (1):
- US Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Ferrando AA, Chinkes DL, Wolf SE, Matin S, Herndon DN, Wolfe RR. A submaximal dose of insulin promotes net skeletal muscle protein synthesis in patients with severe burns. Ann Surg. 1999 Jan;229(1):11-8. doi: 10.1097/00000658-199901000-00002. PMID 9923795